CLINICAL TRIAL: NCT06915038
Title: Circulating Tumor HPV DNA Driven Adjuvant Treatment Deintensification After Transoral Surgery for HPV-Positive Squamous Cell Carcinoma of the Oropharynx
Brief Title: ctHPVDNA in HPV Positive Squamous Cell Carcinoma of the Oropharynx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Michael W. Sim, Associate Professor, Department of Otolaryngology-Head & Neck Surgery, Indiana University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-0895
Record Dates: First submitted 2025-04-01; First posted 2025-04-07 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Squamous Cell Carcinoma of Oropharynx; HPV Positive Cancer; Throat Cancer; Tonsil Cancer
Keywords: NavDX; HPVctDNA; HPV; transoral surgery
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Tonsillar Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Observation (Experimental): Subjects with undetectable postoperative ctHPVDNA levels and either 4 or fewer nodes will have no further adjuvant treatment.
  Interventions: Diagnostic Test: NavDx
- Adjuvant Radiation 30 Gray (Experimental): Subjects with undetectable postoperative ctHPVDNA levels after surgery, negative margins, and five or more positive nodes; or confirmed extranodal extension (ENE) (greater than 2 mm) will undergo deintensified radiation treatment of 30 gray.
  Interventions: Diagnostic Test: NavDx; Radiation: Adjuvant Radiation 30 Gray
- Adjuvant Radiation 40 Gray (Experimental): Subjects with positive postoperative ctHPVDNA will undergo reimaging to evaluate for potentially operable disease, followed by appropriate surgery as indicated. If surgery is performed, repeat ctHPVDNA levels will be checked, and if then negative, subject will be placed in observation or 30 Gy of radiation depending on nodal status.
  If repeat ctHPVDNA level is positive, or subject has no obvious operable disease then subject will undergo 40 Gy of radiation.
  Interventions: Diagnostic Test: NavDx; Radiation: Adjuvant Radiation 40 Gray

INTERVENTIONS:
Diagnostic Test: NavDx — NavDx is a clinically validated blood test to detect circulating tumor HPV DNA (ctHPVDNA). In this study, ctHPVDNA results, in conjuction with specimen analysis, will be used to assign post-surgical adjuvant treatment.
Radiation: Adjuvant Radiation 30 Gray — If undetectable postoperative ctHPVDNA levels and five or more positive nodes, or confirmed extranodal extension (ENE) (greater than 2 mm) deintensified radiation treatment of 30 gray.
  Arms: Adjuvant Radiation 30 Gray
Radiation: Adjuvant Radiation 40 Gray — If detectable postoperative ctHPVDNA, then reimage to evaluate for potentially operable disease, followed by appropriate surgery as indicated. If surgery is performed, repeat ctHPVDNA levels will be checked, and if then negative, subject will be placed in observation if N0 or N1 disease, and 30 Gy of radiation if N2 disease on final pathologic staging. If repeat ctHPVDNA level is positive, or shows no obvious operable disease, then subject will undergo 40 Gy of radiation.
  Arms: Adjuvant Radiation 40 Gray

SUMMARY:
This study is a prospective phase II trial, designed to assess the efficacy and feasibility of adjuvant treatment deintensification guided by ctHPVDNA levels for patients with HPV+OPSCC who undergo transoral surgery and neck dissection.

DETAILED DESCRIPTION:
Oropharyngeal squamous cell carcinoma (OPSCC), commonly known as throat cancer or tonsil cancer, has seen a dramatic rise in incidence over the last twenty years due to the increased incidence of human papillomavirus-positive (HPV) infection and * malignancy within the oropharynx.

The prevailing treatment philosophy within head and neck oncology is that deintensifying treatment could still provide equivalent oncologic outcomes, while further lowering toxicity profiles and improving functional outcomes to minimize the morbidity incurred by patients.

The next frontier in the treatment of HPV+ OPSCC, then, is the potential use of ctHPVDNA in the treatment personalization. Patients could be stratified into risk categories based on their ctHPVDNA levels, and in turn, receive a tailored treatment intensity accordingly.

The goal of this research study is to see if de-intensifying (stopping or scaling back) treatment still provides the same, or perhaps even better, results when compared to standard treatment when using your ctHPVDNA test results as a guide for your treatment.

ELIGIBILITY:
Inclusion Criteria:

Pre-Surgery

* Subjects ≥ 18 years old at the time of informed consent.
* Ability to provide written informed consent and HIPAA authorization.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Primary tumor of the oropharynx (palatine tonsil, tongue base, soft palate, lateral or posterior walls of oropharynx).
* Histopathologically confirmed squamous cell carcinoma.
* Detectable ctHPVDNA from blood samples collected prior to treatment.
* Resectable and accessible tumor with high probability of achieving negative margins.
* Smokers and non-smokers included.
* Tumor stage (AJCC 8th edition): T1 or T2, and select T3 tumors that are mobile and do not invade the larynx.
* Nodal stage (AJCC 8th edition): N0, N1 or N2.
* Mobile neck nodes on physical exam if N positive.
* HPV+ tumor, as determined by p16, in-situ hybridization, real-time polymerase chain reaction, or ctHPVDNA.

Post-Surgery

• Subjects with unknown primaries included if primary is definitively identified and resectable with negative margins or if the palatine and lingual tonsils are thoroughly resected and pathologically proven to be negative for a primary.

Exclusion Criteria:

* Serious medical condition preventing general anesthesia for surgery.
* History of previous head and neck radiation or previous head and neck cancer within 3 years.
* Distant metastatic disease present.
* Subjects with synchronous HPV+ oropharynx primaries
* Prior invasive malignant disease within 3 years, with the exception of non-melanoma skin cancer and thyroid cancer, unless patient is deemed cured or disease free, in which case patient may be included in the study.
* Lactating or pregnant women. Women of childbearing potential must have a negative pregnancy test on the day of surgery. Women are considered to have childbearing potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) unless they meet one of the following criteria:

  1. Has undergone a hysterectomy or bilateral oophorectomy; or
  2. Has been naturally amenorrheic for at least 12 consecutive months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | Up to 24 months post initial surgery
  Time from surgery to first disease recurrence or death from any cause

SECONDARY OUTCOMES:
Local-reginal Control | Up to 24 months post initial surgery
  Number of subjects with no recurrence at primary oropharyngeal site or in the neck nodal basins
Overall Survival | Up to 24 months post initial surgery
  Time from surgery to death from any cause
Distant metastasis rates | Up to 24 months post initial surgery
  Assessed by tissue diagnosis or radiographically of recurrent disease at sites away from the primary tumor and neck nodal basins
Adverse Events | up to 6 months post initial surgery
  Number of subjects that experience adverse events, grades 1-5, as assessed by the National Cancer Institute Common Toxicity Criteria (NCI-CTCAE) version 5.0
Swallowing-related Quality Of Life | 3 months, 6 months, 12 months, and 24 months post initial surgery
  Assessed using MD Anderson Dysphagia Inventory (MDADI)
Gastrostomy tube dependence rates | 12 and 24 months post intial surgery
  Assessed by confirmation of feeding tube in-situ in subject and being utilized for nutrition

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sim, MD, Principal Investigator — Indiana University Melvin and Bren Simon Comprehensive Cancer Center
Locations (2):
- United States (2):
  - IU Health Joe and Shelly Schwarz Cancer Center, Carmel, Indiana
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana